CLINICAL TRIAL: NCT04651283
Title: Effect of Using Adaptive Seating Equipment on Grasping and Visual Motor Integration in Children With Hemiparetic Cerebral Palsy
Brief Title: Effect of Using Adaptive Seating Equipment on Hand Function
Acronym: hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Elsayed Abbass, Mai Elsayed Abbass, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC\012\001765
Record Dates: First submitted 2020-11-16; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: study group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive seating equipment group (Experimental): Study group who received the same selected program for hand function on adaptive swiss ball seating
  Interventions: Other: Adaptive seating equipment group
- Traditional seat group (Active Comparator): Control group who received a specially selected physical therapy program for hand function on a standard chair seating.
  Interventions: Other: Traditional seat group

INTERVENTIONS:
Other: Traditional seat group — Each child in the control group was asked to conduct or follow instructions given for him or her to conduct the following hand function tasks for three successive months of treatment, three times per week (every other day):
  1. Building towers and shapes with different textures weights and bright colors.
  2. Inserting different shapes in the correct hole.
  3. Dropping pellets.
  4. Stringing beads.
  5. Copying square and triangle.
  6. Opening the bottle and close it.
  7. Folding and Crumpling paper.
  8. Cutting paper by scissors.
  9. Tracing line and connecting dots.
  10. Reaching above the level of shoulder.
  11. Reaching across the midline.
  12. Squeezing water out of a sponge.
  13. Buttoning and unbuttoning button.
  14. Playing clapping games.
  15. Turning pages in a book.
  16. Lacing string.
  17. Picking up a small piece of food and bringing it into the palm.
  18. Moving a penny from the palm to the fingers.
  19. Removing socks.
  20. Brush the teeth.
  Other Names: Occupational therapy program for upper limb while the child sitting on chair
  Arms: Traditional seat group
Other: Adaptive seating equipment group — Each child in the study group was asked to conduct or follow instructions given for him or her to conduct the following hand function tasks for three successive months of treatment, three times per week (every other day):
  1. Building towers and shapes with different textures weights and bright colors.
  2. Inserting different shapes in the correct hole.
  3. Dropping pellets.
  4. Stringing beads.
  5. Copying square and triangle.
  6. Opening the bottle and close it.
  7. Folding and Crumpling paper.
  8. Cutting paper by scissors.
  9. Tracing line and connecting dots.
  10. Reaching above the level of shoulder.
  11. Reaching across the midline.
  12. Squeezing water out of a sponge.
  13. Buttoning and unbuttoning button.
  14. Playing clapping games.
  15. Turning pages in a book.
  16. Lacing string.
  17. Picking up a small piece of food and bringing it into the palm.
  18. Moving a penny from the palm to the fingers.
  19. Removing socks.
  20. Brush the teeth.
  Other Names: Occupational therapy program for upper limb while the child sitting on adaptive seating equipment ( swiss ball)
  Arms: Adaptive seating equipment group

SUMMARY:
Objective: The purpose of this study was to evaluate the effect of adaptive swiss ball seating as an alternative for standard chair seating on hand function in children with hemiparesis. Subjects: A total of 30 spastic hemiparetic cerebral palsied children (19 boys and 11 girls), aged 3-6 years participated in this study. They were randomly assigned into control and study groups of equal numbers each consisted of fifteen children (n=15). Methods: Peabody Developmental Motor Scales 2 (PDMS-2) was used to evaluate each child individually before and after three successive months of treatment (3 sessions per week), to assess 2 subtests (the grasping skills and visual motor integration skills) for all children of both groups. Control group who received a specially selected physical therapy program for hand function on a standard chair seating. Study group who received the same selected program for hand function on adaptive swiss ball seating.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of adaptive swiss ball seating as an alternative for standard chair seating on hand function in children with hemiparesis.

In this study, a total of 30 spastic hemiparetic cerebral palsied children (19 boys and 11 girls) aged 3-6 years, they were selected from general hospitals and private centers in kafr El-Sheikh government, randomly assigned to either the control group (n=15), who received a specially selected physical therapy program for hand function on standard chair seating, or the study group (n=15), who received the same selected program for hand function but on adaptive Swiss ball seating. Both groups received 3 sessions per week for 3 successive months. Peabody Developmental Motor Scales 2 (PDMS-2) was used to evaluate each child individually before and after three successive months of treatment, to assess 2 subtests (grasping skills and visual motor integration skills).

ELIGIBILITY:
Inclusion Criteria:

* Children with hemiparetic cerebral palsy.
* The age of the selected children ranged from 3 to 6 years old.
* Degree of spasticity ranged from 1 to 1+, according to Modified Ashworth' Scale (Bohannon and Smith, 1987)
* They were able to follow instructions and understand commands included in both assessment and training procedures.
* They were able to sit independent with trunk control.

Exclusion Criteria:

* Children exposed to orthopedic surgeries or potolinium toxins injection in the last 6 mounth before intervention.
* Children with fixed upper limb deformities
* Children with hearing or visual impairments.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
change is being assessed in grasping score | Change from Baseline grasping score assessed at 3 months
  Assessment of grasping using Peabody Developmental Motor Scale 2 the higher score means a better outcome
change is being assessed in visual motor integration score | Change from Baseline visual motor integration score assessed at 3 months
  Assessment of visual motor integration using Peabody Developmental Motor Scale 2 the higher score means a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Mai Abbass, Ph.D., Study Director — Cairo University; Ahmed Mahrous, Msc, Principal Investigator — Cairo University; Elham Salem, Ph.D., Study Chair — Cairo University
Locations (1):
- Faculty of physical therapy, Cairo university, Cairo, Egypt